CLINICAL TRIAL: NCT01564758
Title: Post Marketing Surveillance on the Efficacy, Safety and Tolerability of Linezolid (Zyvox) in the Treatment of Gram Positive Infections
Brief Title: Post Marketing Surveillance Study on Linezolid
Acronym: A5951090
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5951090; GRAM POSITIVE INFECTIONS
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Results first posted 2012-08-06 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-06

CONDITIONS: Gram-Positive Bacterial Infections
Keywords: non-interventional; non-comparative; open-label study; safety; Linezolid; gram positive infections; Filipino
MeSH Terms: conditions — Gram-Positive Bacterial Infections | interventions — Linezolid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Subjects that are diagnosed with gram positive infection
  Interventions: Drug: Linezolid

INTERVENTIONS:
Drug: Linezolid — 1. Vancomycin-resistant, E. faecium, including concurrent bacteremia: Linezolid for 600mg (IV or oral) every 12 hours for 14-28 days
  2. Nosocomial infection, cSSTI: Linezolid for 600mg (IV or oral) every 12 hours for 10-14 days
  3. Uncomplicated SSTI: Linezolid for 400mg oral every 12 hours for 10-14 days

SUMMARY:
The purpose of this study is to determine if Linezolid is safe for adult Filipino patients diagnosed with gram positive infections.

DETAILED DESCRIPTION:
The subjects were identified after the physician decided to prescribed the drug to the subject.

ELIGIBILITY:
Inclusion Criteria:

* Has clinical diagnosis of of the following, including cases with concurrent bacteremia, when suspected or known to be caused by susceptible strains of anaerobic or aerobic gram positive microorganisms - nosocomial pneumonia, community acquired pneumonia, complicated skin and skin structure infections, uncomplicated skin and skin structure infection, and vancomycin-resistant E. faecium
* Male or female, 18 years old and above

Exclusion Criteria:

* Known hypersensitivity
* Subjects diagnosed with pure gram-negative infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, Filipino patients diagnosed with gram positive infection
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2004-02; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5951090&StudyName=Post%20Marketing%20Surveillance%20study%20on%20Linezolid%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Linezolid: Linezolid (Zyvox) 600 milligram (mg) either intravenously or orally every 12 hours (hrs) for 10 to 28 days or 400 mg orally every 12 hrs for 10 to 14 days until the infection was completely resolved or in accordance with investigator's discretion.
Period: Overall Study
Arm/Group | Linezolid
Started | 99
Completed | 85
Not Completed | 14
Not completed — Death | 8
Not completed — Adverse Event | 3
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Arm/Group | Linezolid
Number analyzed (Participants) | 99
Age Continuous [Mean (Standard Deviation); unit: years] | 59.7 (18.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Any untoward medical occurrence in a participant who received study treatment was considered an AE without regard to possibility of causal relationship.
Time Frame: Baseline up to End of Treatment (EOT) (Day 10 up to 28)
Population: Safety analysis set included all the participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Linezolid
Number analyzed (Participants) | 99
participants | 15

2. Secondary Outcome: Number of Participants With Clinical Response
Description: Clinical response assessed by Investigator at EOT visit as Cure: complete resolution of signs or symptoms of infection and no need to start another antibiotic. Improvement: incomplete resolution of signs or symptoms of infection but no need to start another antibiotic. Failure: death, or need to start another antibiotic. For participants previously assessed as failures, the outcome was failure at subsequent time points.
Time Frame: EOT (Day 10 up to 28)
Population: Efficacy was evaluated for the safety analysis set which included all the participants who received at least 1 dose of study medication
Measure: Number; unit: participants
Arm/Group | Linezolid
Number analyzed (Participants) | 99
participants
  Cure | 57
  Improvement | 31
  Failure | 11

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Linezolid
Serious Adverse Events (participants affected / at risk) | 10/99
Other Adverse Events (participants affected / at risk) | 5/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Linezolid (N=99)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Ill-defined disorder (General disorders) | 3
Septic shock (Infections and infestations) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Linezolid (N=99)
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Protocol did not indicate primary or secondary endpoints and all determination of primary or secondary endpoints were arbitrary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.